CLINICAL TRIAL: NCT07226193
Title: Pulse Arrival Time as an Alternative Biomarker to Detect Lower-Extremity Peripheral Artery Disease
Brief Title: Detecting Peripheral Artery Disease With the Pulse
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0685-25-EP
Record Dates: First submitted 2025-10-30; First posted 2025-11-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Peripheral Artery Disease (PAD)
Keywords: pulse arrival time; atherosclerosis; peripheral artery disease; portable peripheral artery disease detection
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis

STUDY DESIGN:
Intervention Model Description: To address the objective of Specific Aim #1 & #2, two groups of participants are defined as needing to complete the study: 1) patients with peripheral artery disease and 2) age-matched controls. All participants will participate in a single laboratory visit where 1) the experimental device will be tested, 2) an ankle-brachial index will be performed, and 3) a 6-min walking test will be performed.
  To address the objectives of Specific Aim #3, two groups of participants are defined as needing to complete the study: 1) younger adults (19-54 yrs) and 2) older adults (+55 yrs). All participants will participate in a single laboratory visit where 1) the experimental device will be tested, 2) an ankle-brachial index will be performed, and 3) a 6-min walking test will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Laboratory Visit #1 (Experimental): During the first and only laboratory visit, subjects will be tested 1) with the experimental device, 2) an ankle-brachial index will be performed, and 3) a 6-min walking test will be performed.
  Interventions: Device: Segmental pulse arrival time assessment

INTERVENTIONS:
Device: Segmental pulse arrival time assessment — A proprietary device has been developed to obtain segmental pulse arrival times in the arms and legs. Using this information, the propagation time of the pulse is being investigated as a biomarker to detect the presence of lower-extremity atherosclerosis. Furthermore, the impacts of aging on the biomarker will be assessed.

SUMMARY:
1) The purpose of this study is to assess segmental pulse arrival time (PAT) as an alternative biomarker to detect lower-extremity peripheral artery disease (PAD), and to investigate the impacts of local skin heating and foot elevation. The secondary purpose will be to investigate the impacts of age on segmental PAT. The subject population will include any adults 19 years of age or older with or without PAD. Exclusion criteria include having an aortic aneurysm with or without previous intervention, previous revascularization surgeries of the arteries in the legs/aorta, walking impairments independent of PAD, gangrene or ulcers of the toes/feet, and currently pregnant or breastfeeding. 3) All aims of the present study will be completed with a single laboratory visit. Descriptive measurements will include height, weight, age, sex, body fat percentage, and self-reported medication and health history. Subjects will lie in the supine position for 20-min. After rest, either the ankle-brachial index (ABI) or PAT will be assessed. After 10-min of further rest, the other measurement will be performed. ABIs will be assessed according to current guidelines: blood pressures will be assessed in the dorsal pedis and tibialis posterior arteries of both legs and the brachial arteries of both arms using a blood pressure cuff and Doppler ultrasound. PAT will be simultaneously assessed in both arms and legs using an investigational device with a 3-lead electrocardiogram sensor and four photoplethysmography (PPG) sensors. A PPG sensor will be applied to both middle fingers and both big toes. Signals will be collected for 15-min with finger and toe sensor temperatures at 30 C. Toe sensor temperature will then be elevated to 45 C for 15-min. Finally, toe sensor temperature will remain at 45 C, and the feet will be elevated 8-in with a soft cushion for 15-min. Blood pressure in the foot will be assessed before and after foot elevation with Doppler ultrasound. Thermal images of the fingers and toes will be assessed before and after using the investigational device. Subjects will then participate in a 6-min walking test (6MWT) to objectively establish walking capacity. The 6MWT will be performed in accordance with current guidelines. Segmental PATs will be compared with ABI and 6-min walking time to determine if segmental PATs can predict lower-extremity PAD (ABI) and the associated walking impairment (6MWT). This study is expected to last ~2.5hrs. 4) There will be no follow-up.

DETAILED DESCRIPTION:
Specific Aim 1: Determine if segmental pulse arrival times can predict lower-extremity peripheral artery disease assessed with ankle-brachial index and the 6-min walking test.

Specific Aim 2: Determine if local skin heating of the toes and foot elevation improves the prediction of peripheral artery disease using segmental pulse arrival times.

Specific Aim 3: Determine the effects of age on segmental pulse arrival times.

After the process of informed consent, descriptive measurements will be assessed. Descriptive measures include height, weight, body composition, age, and sex. Height and weight will be assessed with a standard stadiometer and scale, respectively. Body composition will be assessed non-invasively with bio-electric impedance analysis (Omron HBF-306C Handheld Scanner, OMRON Healthcare, Kyoto, Japan). Bioelectric impedance devices send a small electric current through the body and estimates body fat percentage based on the impedance to electrical flow through the body segments. Our bio-electric impedance device creates a circuit between the hands and feet of the subject to estimate body fat percentage. The electric current used in bioelectric impedance devices is very small and cannot be felt by the participant. Subjects will also self-report their medication and health history.

After the assessment of descriptive measurements, subjects will rest in the supine position for 20-min. After 20-min of rest, the subjects will have either ankle-brachial index (ABI) or segmental pulse arrival times (PATs) assessed. After a 10-min period of rest, the other measurement will be assessed (either ABI or PAT). The order of ABI and PAT will be randomized, and all subjects will have ABI and PAT assessed.

1a) Assessment of PAT with the Investigational Device: The subjects will be instrumented with an investigational device comprised of an array of four photoplethysmography (PPG) sensors and one 3-lead electrocardiogram (ECG) sensor. Electrocardiogram is a non-invasive technique that is used to monitor the electrical dipoles generated by membrane potentials within the myocardium and electrical conduction systems of the heart. PPG is a non-invasive technique to assess hemoglobin content within the microcirculation of the skin. Our PPG sensors are applied superficially on the skin and shines continuous-intensity green light into the skin (580 nm). The green light is absorbed by hemoglobin. Therefore, by the modified Beer-Lambert principle, the amount of light reflected back to the PPG unit gives an index of hemoglobin content within the microvasculature. The PPG and ECG sensors are integrated into a microcontroller (small computer), which reads the voltages of the sensors and displays the data in real time in a custom computer software. Each PPG sensor will have a skin-safe double-sided adhesive attached to the sensor housing. Two PPG sensors will be adhered to both middle fingers on the palmar side of the hands. Two PPG sensors will be adhered to the plantar aspect of both big toes. Altogether, there will be one PPG sensor per hand and one PPG sensor per foot. The ECG sensor will be applied to form limb leads: one electrode per wrist on the ventral aspect of the forearm and one electrode on a hair-free portion of the left leg. If an adequate ECG signal is not obtained using limb leads, then chest leads will be utilized. In this configuration, electrodes will be placed inferior to the left and right clavicle, and medial to the shoulders, and one electrode will be placed on the left lateral aspect of the ribcage near the apex of the heart. Once all sensors have been placed, the subject will rest in the supine position. Blood pressure will be assessed in the arm with a standard automatic blood pressure device. Systolic blood pressure in the foot will be assessed with Doppler ultrasound on the dorsal pedis artery and a standard blood pressure cuff around the lower leg. Next, the temperature of the sensor housings attached to the fingers and toes will be warmed to 30 C, which is thermoneutral with skin temperature. After 15-min of signal collection, the toe sensor housings will be heated to 45 C to warm up the skin of the toes, and the finger sensor housings will remain warmed at 30 C. After 15-min of additional signal collection, the lower legs will be elevated 8-in with a soft cushion. The toe sensors will remain heated at 45 C, and the finger sensors will remain at 30 C. Signals will be collected continuously for an additional 15-min. Finally, systolic blood pressure in the foot during elevation will be assessed with Doppler ultrasound on the dorsal pedis artery and a standard blood pressure cuff around the lower leg. For all conditions, PAT will be calculated for each arm and each leg as the difference in time between the R-wave appearing in the ECG signal and the pulse wave appearing in the distal PPG signals. All four PAT values will be used to develop a composite score to estimate the presence of lower-extremity PAD. Leg asymmetry will be assessed with the ratio of PATs from left and right legs. Atherosclerotic plaque-mediated pulse wave slowing will be assessed as the ratio of PATs in the arms compared to the legs. The product of these ratios forms the composite score to detect lower-extremity PAD, which is sensitive to both 1) asymmetry in PATs in the legs (may indicate unilateral lower-extremity PAD) and 2) longer PATs in the legs compared to the arms (may indicate the presence of lower-extremity PAD).

1b) Thermal Imaging: Immediately prior to applying and immediately after removing the PPG sensors, a thermal imaging camera (FLIR T540) will be used to take a thermal image of the skin where the PPG sensors will be/were applied. Thermal images will be taken after warming to 30 C and 45 C. The purpose of using the thermal camera is to document the local skin temperature before and after using the investigational device. The thermal camera will automatically select the warmest region of the image and document the temperature. Of note, the thermal imaging camera will be zoomed in on the fingers and toes where the PPG sensors were located, and no identifiable body parts (e.g., face) or clusters of body parts (e.g., zoomed out images) will be included in the thermal images. Therefore, the risk of identifying subjects with the thermal images will be minimized.

2) Assessment of ABI: ABI will be assessed according to current guidelines established by the American Heart Association and the American College of Cardiology. Blood pressures will be assessed in both legs and in both arms. For all blood pressure assessments, the blood pressure cuff will be manually inflated to a supra-systolic pressure. During slow manual cuff deflation, a Doppler ultrasound (non-invasive) will be used to listen for the first Korotkoff sound, which is the systolic blood pressure. Using this procedure, the systolic blood pressure will be quantified for both the ipsilateral dorsalis pedis and posterior tibial arteries for both legs. Furthermore, systolic blood pressure will be assessed in the brachial arteries of both arms. ABI will be quantified as the ratio of the higher systolic blood pressure in the legs divided by the higher systolic blood pressure in the arms.

3) 6-minute walking test: After the assessments of ABI and PAT, subjects will participate in a 6-min walking test to objectively quantify exercise capacity. Two cones will be separated by 30 m on a straight and flat walkway. Subjects will be instructed to walk back and forth between the cones as fast as they can for 6-min to achieve the farthest distance that they can. Subjects will be allowed to rest during the test, but the stopwatch time will not be stopped. All components of the test will be explained clearly prior to performing the test. Comprehension of the objectives of the test will be confirmed prior to initiating the test. Prior to performing the 6-min walking test, blood pressure, heart rate, and the rating of perceived exertion (RPE) will be recorded in the seated position. Furthermore, blood pressure, heart rate, and RPE will be recorded with the subject in the seated position immediately after exercise and every 5-min thereafter until the pre-exercise heart rate and blood pressure are re-established (w/in +/-5 beats and +/-5 mmHg) in alignment with American College of Sports Medicine guidelines.

The study duration is expected to be ~2.5 hrs, and there will be no follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. be able to provide written informed consent
2. be 19 years of age or older
3. having or not having a diagnosis of peripheral artery disease

Exclusion Criteria:

1. having a current or pervious aortic aneurysm with or without previous intervention
2. having previous revascularization surgeries (open or endovascular) of the legs or aorta
3. having walking impairments independent of lower-limb ischemia (e.g., musculoskeletal injury)
4. having gangrene or ulcers of the toes/feet
5. being currently pregnant or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-05 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Segmental pulse arrival times | Day 1
  Pulse arrival time will be assessed in both arms and legs with the investigational device
Ankle-brachial index | Day 1
  Segmental blood pressures in the arms and ankles will be assessed as an index of the presence and/or severity of lower-extremity atherosclerosis. The ankle-brachial index is the standard screening assessment for peripheral artery disease in the lower-extremities.
6-min walking distance | Day 1
  The 6-min walking test is a standard assessment of mobility in older adults and in patients with peripheral artery disease. The 6-min walking test will be performed to quantify the level of walking impairment in patients with peripheral artery disease.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nebraska at Omaha Health Science Collaborative, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD will be shared upon request to journals for the purpose of publication. Specific IPD will include the primary outcome measures of this study.